CLINICAL TRIAL: NCT02962986
Title: A Comparison of Intermittent Intravenous Boluses of Phenylephrine and Norepinephrine to Prevent Spinal-induced Hypotension in Cesarean Deliveries: a Randomized Controlled Study
Brief Title: A Comparison of Intermittent Intravenous Boluses of Phenylephrine and Norepinephrine to Prevent Spinal-induced Hypotension in Cesarean Deliveries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-07
Record Dates: First submitted 2016-11-07; First posted 2016-11-15 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Hypotension
Keywords: vasopressor; blood pressure; cesarean section; spinal anesthesia
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- norepinephrine 6mcg (Active Comparator): norepinephrine, given as 1mL IV boluses, to treat post-spinal hypotension
  Interventions: Drug: Norepinephrine
- phenylephrine 100mcg (Active Comparator): phenylephrine, given as 1mL IV boluses, to treat post-spinal hypotension
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Norepinephrine — Norepinephrine diluted in 5% dextrose solution to a concentration of 6mcg/mL
  Other Names: Norepinephrine bitartrate
  Arms: norepinephrine 6mcg
Drug: Phenylephrine — Phenylephrine diluted in 0.9% normal saline solution to a concentration of 100mcg/mL
  Other Names: Phenylephrine Hydrochloride
  Arms: phenylephrine 100mcg

SUMMARY:
Hypotension is a very common complication of spinal anesthesia for cesarean delivery, and can have unwanted side effects on both mother and fetus if not treated promptly. Phenylephrine has been the drug of choice to treat this spinal-induced hypotension. Although phenylephrine is safe to use for this indication, it has been associated with reflex bradycardia and a reduction in cardiac output.

Norepinephrine is a potent vasopressor used to treat hypotension in the critical care setting. Recent studies have looked at norepinephrine's use in the obstetric setting, and have shown that it can be used safely and also has favourable hemodynamic properties when compared to phenylephrine, with less bradycardia and less depression of cardiac output.

The investigators recently conducted a study to determine the ED90 of norepinephrine, and now plan to compare bolus doses of phenylephrine to norepinephrine for treating hypotension following spinal anesthesia for cesarean section.

The investigators hypothesize that norepinephrine, when given as a bolus to prevent post spinal hypotension, will result in around 70% relative decrease in the rate of bradycardia when compared to phenylephrine in patients undergoing elective cesarean delivery under spinal anesthesia.

DETAILED DESCRIPTION:
Norepinephrine is a potent vasopressor used to treat hypotension in the critical care setting. Recent studies have looked at norepinephrine's use in the obstetric setting, and have shown that it can be used safely and also has favourable hemodynamic properties when compared to phenylephrine, with less bradycardia and less depression of cardiac output. These studies have been limited to using norepinephrine as an infusion and there is limited data with it being used as a bolus to prevent hypotension. A recent study was undertaken at Mount Sinai hospital to determine the ED90 of norepinephrine to treat post spinal hypotension. Secondary outcome data from this trial showed that the incidence of bradycardia associated with this treatment is approximately 7.5%, several times less when compared to the reported 30% with phenylephrine. It would therefore be prudent at this stage to undertake a randomized trial comparing the hemodynamic profile of phenylephrine (our standard practice) and norepinephrine used as intermittent boluses to prevent hypotension and avoid decrease in heart rate during cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Elective CS under spinal anesthesia
* Normal singleton pregnancy beyond 36 weeks gestation
* ASA physical status 2-3
* Current (pregnant) weight 50-100 kg, height 150-180 cm
* Age over 18 years

Exclusion Criteria:

* Patient refusal
* Inability to communicate in English
* Allergy or hypersensitivity to phenylephrine
* Preexisting or pregnancy-induced hypertension
* Cardiovascular or cerebrovascular disease
* Fetal abnormalities
* History of diabetes, excluding gestational diabetes
* Contra-indications for spinal anesthesia
* Allergy or hypersensitivity to sulfite
* Use of monoamine oxidase inhibitors, triptyline or imipramine antidepressants
* Untreated hyperthyroid patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Bradycardia: Heart rate less than 50 bpm | 30 minutes
  Heart rate less than 50 bpm, from induction of spinal anesthesia

SECONDARY OUTCOMES:
Hypotension: Systolic blood pressure less than 80% of baseline | 30 minutes
  Systolic blood pressure below 80% of baseline, from induction of spinal anesthesia to delivery of the fetus.
Number of hypotensive episodes | 30 minutes
  The number of times the systolic blood pressure measures below 80% of baseline, from induction of spinal anesthesia to delivery of the fetus.
Hypertension: Systolic blood pressure at or above 120% of baseline | 30 minutes
  Systolic blood pressure at or above 120% of baseline, from induction of spinal anesthesia to delivery of the fetus.
Tachycardia: Heart rate greater than 30% of baseline | 30 minutes
  Heart rate greater than 30%, from induction of spinal anesthesia to delivery of the fetus.
Presence of nausea | 30 minutes
  Presence of nausea in patients from induction of spinal anesthesia to delivery of the fetus.
Number of episodes of nausea | 30 minutes
  The number of episodes of nausea experienced by patients from induction of spinal anesthesia to delivery of the fetus.
Presence of vomiting | 30 minutes
  Presence of vomiting in patients from induction of spinal anesthesia to delivery of the fetus.
Number of episodes of vomiting | 30 minutes
  The number of episodes of vomiting experienced by patients from induction of spinal anesthesia to delivery of the fetus.
Total dose of study drug given | 30 minutes
  Total dose of study drug given from induction of spinal anesthesia to delivery of the fetus.
Apgar scores | 1 minute and 5 minutes
  The Apgar scores of the infant at 1 and 5 minutes post delivery.
Umbilical artery pH | 24 hours
  Umbilical artery pH
Umbilical artery partial pressure of carbon dioxide | 24 hours
  Umbilical artery partial pressure of carbon dioxide
Umbilical artery partial pressure of oxygen | 24 hours
  Umbilical artery partial pressure of oxygen
Umbilical artery bicarbonate (mmol/L) | 24 hours
  Umbilical artery bicarbonate
Umbilical artery base excess (mmol/L) | 24 hours
  Umbilical artery base excess
Umbilical vein pH | 24 hours
  Umbilical vein pH
Umbilical vein partial pressure of carbon dioxide | 24 hours
  Umbilical vein partial pressure of carbon dioxide
Umbilical vein partial pressure of oxygen | 24 hours
  Umbilical vein partial pressure of oxygen
Umbilical vein bicarbonate (mmol/L) | 24 hours
  Umbilical vein bicarbonate
Umbilical vein base excess (mmol/L) | 24 hours
  Umbilical vein base excess

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No